CLINICAL TRIAL: NCT05466305
Title: Immunological and Microbiological Assessment of Maxillary Acrylic Resin Complete Dentures Reinforced by Gold Plated Cr-Co Palatal Plate
Brief Title: Assessment of Maxillary Acrylic Resin Complete Dentures Reinforced by Gold Plated Cr-Co Palatal Plate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Shady El Naggar, Clinical Professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01012336911
Record Dates: First submitted 2022-07-08; First posted 2022-07-20 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Denture Stomatitis
Keywords: Gold; Chrome; Denture; Mucosa
MeSH Terms: conditions — Stomatitis, Denture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary complete denture reinforced by chrome cobalt alloy (Placebo Comparator): Completely edentulous patients treated by maxillary complete denture reinforced by chrome cobalt alloy
  Interventions: Device: Gold plated chrome cobalt alloy
- Maxillary complete denture reinforced by gold plated chrome cobalt alloy (Experimental): Completely edentulous patients treated by maxillary complete denture reinforced by gold plated chrome cobalt alloy
  Interventions: Device: Gold plated chrome cobalt alloy

INTERVENTIONS:
Device: Gold plated chrome cobalt alloy — Acrylic resin complete denture having a metal chrome cobalt palatal plate which plated by gold
  Other Names: Completely edentulous patients treated by maxillary complete denture reinforced by gold plated chrome cobalt alloy

SUMMARY:
Gold is widely used in prosthetics. Its use ranges from being employed in the fabrication of removable dentures, where the inner surface permanently touching oral cavity tissues, through to fixed dentures, and even some structures of certain implantological systems. All such items can be made of galvanized gold. Thus, new technologies have made gold and its alloys a kind of a universal material.

DETAILED DESCRIPTION:
Gold is widely used in prosthetics. Its use ranges from being employed in the fabrication of removable dentures, where the inner surface permanently touching oral cavity tissues, through to fixed dentures, and even some structures of certain implantological systems. All such items can be made of galvanized gold. Thus, new technologies have made gold and its alloys a kind of a universal material.

Using metal alloys (gold alloys included) to make the framework for removable dentures is much better than using acrylic resin. This because the alloys have almost no destructive influence over the dentures bearing area. Due to the precise way it is made, the stability of shape, the lack of internal stresses and the close contact with the dentures bearing area, it is possible to achieve very good retention of the denture over a long span of time. Another advantage is that the metal framework conducts temperature changes and this facilitates keeping the tissues in good health. Also, a denture metal framework makes it much easier for the patient to maintain good oral hygiene by lowering the risk of plaque accumulation. However, a metal framework has a disadvantage as well - prosthesis relining cannot be made.

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous maxillary and mandibular ridges
2. Healthy mucosa and absence of remaining roots
3. Good physical and mental health
4. Willing to give informed consent
5. Normal maxilla-mandibular relationship Angle Class I
6. Adequate bone quality and quantity in terms of width and height in the anterior maxillary mandibular ridges verified by preoperative cone beam CT
7. Adequate inter-arch space to accommodate maxillary and mandibular implant prostheses

Exclusion Criteria:

1. Uncontrolled diabetes
2. Smoking habits
3. Radiotherapy
4. Clinical or radiographic signs of pathologic conditions
5. Osteoporosis
6. Patients on corticosteroids
7. Bruxism

Ages: 4 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Immunological assessment using Salivary IgA level through ELISA test | 45 days
  Immunological assessment of maxillary complete denture reinforced by gold plated Cr-Co alloy

SECONDARY OUTCOMES:
Microbiological assessment using Staphylococcus Aureus, Staphylococcus Epidermis and Candida Albicans Colonization | 45 days
  Microbiological assessment of maxillary complete denture reinforced by gold plated Cr-Co alloy

CONTACTS AND LOCATIONS:
Overall Officials: Shady M. El Naggar, PhD, Principal Investigator — Badr University in Cairo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05466305/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05466305/ICF_002.pdf